CLINICAL TRIAL: NCT03320538
Title: Efficacy and Safety of Hou Gu Mi Xi in Patients With Peptic Ulcer Diseases: A Multicenter, Randomized, Double-blinded, Controlled Trial
Brief Title: Efficacy and Safety of Hou Gu Mi Xi in Patients With Peptic Ulcer Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Collaborators: Jiangxi Hospital of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); The Third Affiliated Hospital of Nanchang University (Other); Nanchang Hongdu Hospital of Traditional Chinese Medicine (Unknown); Nanchang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); The Nanchang Third Hospital (Unknown); Xinyu People's Hospital (Unknown); Xinyu Hospital of Traditional Chinese Medicine (Unknown); Jiujiang No.1 People's Hospital (Other); Jiujiang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Xu Zhou, Lecturer, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JXUTCM-EBM-03
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Peptic Ulcer Disease
Keywords: Hou Gu Mi Xi; peptic ulcer disease; traditional Chinese medicine; randomized controlled trial; dietary therapy
MeSH Terms: conditions — Peptic Ulcer | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hou Gu Mi Xi (Experimental): Basic treatment period (0 to 2rd week): Patients with infection of Helicobacter pylori receive rabeprazole (once 20 mg, twice a day), bismuth potassium citrate (once 0.3 g, twice a day), amoxicillin (once 1 mg, twice a day), and furazolidone (once 0.1 g, twice a day), and patients without infection of Helicobacter pylori only receive rabeprazole (once 20 mg, twice a day) and bismuth potassium citrate (once 0.3 g, twice a day).
  Maintain treatment period (3rd to 6th week): Patients in this arm receive Hou Gu Mi Xi (once 10 g, twice a day).
  Recuperation period (7th to 52th week): Patients in this arm receive Hou Gu Mi Xi (once 10 g, twice a day).
  Extensional observational period (53 to 104 weeks): no intervention.
  Interventions: Other: Hou Gu Mi Xi
- Hou Gu Mi Xi + rabeprazole (Experimental): Basic treatment period (0 to 2rd week): Patients with infection of Helicobacter pylori receive rabeprazole (once 20 mg, twice a day), bismuth potassium citrate (once 0.3 g, twice a day), amoxicillin (once 1 mg, twice a day), and furazolidone (once 0.1 g, twice a day), and patients without infection of Helicobacter pylori only receive rabeprazole (once 20 mg, twice a day) and bismuth potassium citrate (once 0.3 g, twice a day).
  Maintain treatment period (3rd to 6th week): Patients in this arm receive Hou Gu Mi Xi (once 10 g, twice a day) plus rabeprazole (once 10 mg, once a day).
  Recuperation period (7th to 52th week): Patients in this arm receive Hou Gu Mi Xi (once 10 g, twice a day).
  Extensional observational period (53 to 104 weeks): no intervention.
  Interventions: Other: Hou Gu Mi Xi; Drug: Rabeprazole
- Placebo + rabeprazole (Placebo Comparator): Basic treatment period (0 to 2rd week): Patients with infection of Helicobacter pylori receive rabeprazole (once 20 mg, twice a day), bismuth potassium citrate (once 0.3 g, twice a day), amoxicillin (once 1 mg, twice a day), and furazolidone (once 0.1 g, twice a day), and patients without infection of Helicobacter pylori only receive rabeprazole (once 20 mg, twice a day) and bismuth potassium citrate (once 0.3 g, twice a day).
  Maintain treatment period (3rd to 6th week): Patients in this arm receive Placebo of Hou Gu Mi Xi (once 10 g, twice a day) plus rabeprazole (10 mg/d, qd).
  Recuperation period (7th to 52th week): Patients in this arm receive Hou Gu Mi Xi (once 10 g, twice a day).
  Extensional observational period (53 to 104 weeks): no intervention.
  Interventions: Other: Placebo; Drug: Rabeprazole
- Placebo (Placebo Comparator): Basic treatment period (0 to 2rd week): Patients with infection of Helicobacter pylori receive rabeprazole (once 20 mg, twice a day), bismuth potassium citrate (once 0.3 g, twice a day), amoxicillin (once 1 mg, twice a day), and furazolidone (once 0.1 g, twice a day), and patients without infection of Helicobacter pylori only receive rabeprazole (once 20 mg, twice a day) and bismuth potassium citrate (once 0.3 g, twice a day).
  Maintain treatment period (3rd to 6th week): Patients in this arm receive placebo of Hou Gu Mi Xi (once 10 g, twice a day).
  Recuperation period (7th to 52th week): Patients in this arm receive Hou Gu Mi Xi (once 10 g, twice a day).
  Extensional observational period (53 to 104 weeks): no intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Hou Gu Mi Xi — Hou Gu Mi Xi is an oatmeal-liked, solid food (dry or dissolved eating).
  Arms: Hou Gu Mi Xi; Hou Gu Mi Xi + rabeprazole
Other: Placebo — The placebo is as same as Hou Gu Mi Xi in respect of color, taste, and smell.
  Arms: Placebo; Placebo + rabeprazole
Drug: Rabeprazole — Rabeprazole is produced by Shanghai Xinyi Pharmaceutical Corp. Ltd.
  Other Names: Trade name: Xin Wei An
  Arms: Hou Gu Mi Xi + rabeprazole; Placebo + rabeprazole

SUMMARY:
This trial aims to determine whether Jiangzhong Hou Gu® Mi Xi™ is an effective intervention to improve symptoms and indicators in patients with spleen qi deficiency and peptic ulcer diseases.

DETAILED DESCRIPTION:
Peptic ulcer diseases (PUD) is a common kind of digestive system disease, which mostly involves in stomach and duodenum. PUD may occur at any age but mainly at 30 to 49 years (the proportion was about 50% among all PUD patients). One epidemiological survey showed that the incidence was 17.2% in China and the ratio of gastric to duodenal ulcer diseases was about 1:2.

The two most common reasons for causing PUD were infection of Helicobacter pylori (Hp) and long-term use of non-steroid anti-inflammatory drug (NSAID). In recent year, the infection rate of Hp increased continuously. Among Chinese PUD patients, 92.6% infected Hp, and 72.2% patients who infected Hp occurred PUD. The typical symptoms of PUD were upper abdominal pain, abdominal distension, nausea and vomiting, belching, and inappetence. These symptoms were cyclical, rhythmic and chronic, and were usually tolerable. However, PUD may progress to bleeding or perforation, and these acute complication always lead to worse prognosis.

Along with the development of medical science, traditional Chinese medicine (TCM) is playing an increasingly rule in treatment of PUD. Shen Ling Bai Zhu San is a classic Chinese medicinal formulae originally described in Tai Ping Hui Min He Ji Ju Fang in the Fang Song Dynasty (1102 AD), which is composed of ginseng, tuckahoe, atractylodes, baked licorice, coixenolide, Chinese yam, lotus seed, shrinkage fructus amomi, platycodon grandiflorum, white hyacinth bean, and dried orange peel. It is mainly used for treating the syndrome of spleen qi deficiency, including dyspepsia, chest and stomach distress, borborygmus and diarrhea, limb weakness, thin body, sallow complexion, pale tongue with white and greasy coating, and weak and slow pulse, etc.

In the theory of TCM, spleen is the source for producing qi and blood and thus is the root of life. PUD are classed as the syndrome of "Pi Man (fullness)" in TCM, which was caused by spleen qi deficiency, imbalance of rise and fall, and/or stagnation of qi activity. Shen Ling Bai Zhu San could invigorate spleen by supplying spleen and remove wet, nourish the stomach and intestine, and thus improve symptoms of PUD. Pharmacological researches showed that Shen Ling Bai Zhu San could regulate function of anaerobic and aerobic bacteria in gastrointestinal tract; specifically, it could promote growth of probiotics (e.g. bifidobacterium) and inhibit main drug-resistant strains (e.g. enterococcus), and thereby enhance the body's self-healing function of ulcer.

Jiangzhong Hou Gu® Mi Xi™ is a dietary therapy form of Shen Ling Bai Zhu San, of which removes atractylodes and platycodon grandiflorum (two herbs that could not be used as food) from Shen Ling Bai Zhu San, and adds perilla leaf for adapting a dietary therapy. Jiangzhong Hou Gu® Mi Xi™ used the main formula of Shen Ling Bai Zhu San, so that it could theoretically maintain the treatment effects. Although the reliable health effects of Shen Ling Bai Zhu San has been proved in previous studies, Jiangzhong Hou Gu® Mi Xi™ is optimized in formula and its preparations changed from electuary to rice paste, so that its functional mechanism and efficacy may also be different. Therefore, the investigators plan to perform a hospital-based randomized controlled trial, enroll patients from 13 hospitals in Jiangxi Province in China, aims to assess function and safety of Jiangzhong Hou Gu® Mi Xi™ in patients with spleen qi deficiency and PUD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should be diagnosed as gastric or duodenal ulcer under endoscope; the diameter of ulcers range from 0.3 to 1.0 cm; no indicator of bleeding or perforation.
2. Patient should be diagnosed as syndrome of spleen qi deficiency, that is, meet 2 main symptoms of spleen deficiency and 2 main symptoms of qi deficiency, or have 2 main symptoms of spleen deficiency, 1 main symptoms of qi deficiency and tongue symptoms as follow:

   * Main symptoms of spleen deficiency: a) poor appetite; b) abnormal stool (loose, diarrhea); c) abdominal distention after meal or at afternoon
   * Main symptoms of qi deficiency: a) fatigue and weak; b) tired mind and taciturnity
   * Secondary symptoms: a) tastelessness, hypodipsia, like hot drink, or polysialia; b) abdominal pain, as a result either patients like warm or press; pain remits after meal or occurs when work; c) nausea and vomiting; d) tightness in stomach; e) abnormal bowel sounds; f) lean or puffiness; g) sallow complexion; h) powerless defecation weakness; i) edema
   * Tongue symptoms: pale or swollen or teeth-printed tongue with thin and white fur
3. Age is between 18 to 70 years
4. Sign the informed consent

Exclusion Criteria:

1. Patients who have complex peptic ulcer (i.e. have gastric and duodenal ulcer meanwhile)
2. Patients who have history of ulcer complications (e.g. bleeding or perforation)
3. Patients who have indicators of ulcer complications, including bleeding (Forrest stage I, IIa and IIb) or perforation (area of ulcer is more than 1 cm).
4. Patients whose ulcer have healed, that is, the ulcer is at healing stage or scarring stage according to the diagnosis criteria in Consensus View of Integrated Chinese and Western Medicine on Diagnosis and Treatment of Peptic Ulcer (2011, Tianjin)
5. Patients who took proton-pump inhibitor more than 3 days within 15 days, or took non-steroid anti-inflammatory drugs for a long term
6. Female patients who are pregnant or breast-feeding, or prepare to pregnant for pregnancy within 2 years
7. Patients who are allergic to sample or sample composition
8. Patients who are allergic to sample or sample composition
9. Patients who have impaired liver function, including one of following condition: a) total bilirubin > 35 μmol/L; b) alanine transaminase >2 upper limit of normal (ULN); or c) aspartate aminotransferase >2 ULN
10. Patients who have impaired kidney function, that is, serum creatinine >2 ULN
11. Patients who have obviously abnormal electrocardiogram
12. Patients who have stool occult blood, that is, positive result in immunoassay or iron elemental test, and the results continue to be positive after 3 days of vegetarian diet.
13. Patients who undertaken drugs that could damage stomach and intestine, or experienced side effects of dyspepsia for undertaking non-steroidal anti-inflammatory drugs, theophylline, oral antibiotic or potassium supplements within 3 months
14. Patients who are receiving any agents or other intervention for treating his/her gastrointestinal disorder
15. Patients with any malignant tumor
16. Patients who have severe mental disorders so that could not control his/her action and coordinate the treatment in this trial.
17. Patients who are unwilling to provider personal information and enter this trial
18. Patients who cannot understand and sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Total effective rate | At baseline, and 12, 26, 52, and 104 weeks
  The ulcer was classified for 6 grades:
  A1: The ulcer is round or elliptical with the center covers thick and white fur; it can be accompanied by errhysis or blood clot, and was surrounded by the obvious flush, hyperemia and edema.
  A2: The ulcer is covered by yellow or white fur, no bleeding, alleviated congestion and edema H1: The ulcer is healing, no hyperemia and edema disappear around the ulcer; the ulcer moss becomes thin, subside, accompanied by the new capillaries.
  H2: The ulcer continuously changes to shallow and small. The surrounding mucosa plica centralized to the ulcer.
  S1: The white fur of ulcer disappears and the new ulcer mucosa presents red. S2: The new ulcer mucosa goes from red to white.
  Clinical cure: The ulcer heals with or without scar Markedly effective: The healing of ulcer reaches grade H2, or improves 2 grades Effective: The healing of ulcer reaches grade H1, or improves 1 grades Non-effective: No efficacy by the endoscopic observation
Quality of ulcer healing | At baseline and 12 and 26 weeks
  According to Pan et al's method, we will classify the quality of ulcer healing as three ranks by histological assessment: 1) good: integral villus and epithelium, many glands, good morphology, many blood capillary, and few inflammatory cells infiltration. 2) fair: short villus, incomplete or rough epithelium, less glands, structural distortion, few blood capillary, and moderate inflammatory cells infiltration; 3) poor: a little new epithelial cell, poor integrity of epithelium, poor morphology of villus and glands, very few blood capillary, and large amount of inflame cells.
Changes in Spleen Qi Deficiency Symptoms Grading and Quantifying Scale (unit: score on a scale) | At basline and 6, 12, 26, 52 and 104 weeks
  This outcome will be assessed based on the Spleen Qi Deficiency Symptoms Grading and Quantifying Scale (SQD scale) score. Construct of SQD scale: A total of 15 items, of which 7 items assess main symptoms, including stomach pain, stomach distension, acid reflux, abdominal distension, powerless defecation, fatigue and weak, and inappetence; 8 items assess secondary symptoms, including stomach tightness, stomach burn, belching, nausea and vomiting, abnormal stool, tired mind and taciturnity, sallow complexion, and tastelessness and hypodipsia.
  Scale ranges and explanations: Assessment of each item includes three aspects: degree, frequency in one day, and episodes within one week. The total score of each item is the sum of points of the three aspects. The higher score indicate the worse symptom. The items for assessing main symptoms are double weighted. The score range is 0 to 283 point.

SECONDARY OUTCOMES:
Ulcer area (cm^2) | At baseline and 12, 26, 52 and 104 weeks
  Ulcer area was measured under endoscope.
Recurrence rate | At baseline and 12, 26, 52 and 104 weeks
  For patients who have cured, ulcer is observed again under endoscope during the follow up period is considered as recurrence.
Eradication rate of helicobacter pylori | At 12, 26, 52 and 104 weeks
  For patients infected with helicobacter pylori, the helicobacter pylori is considered as being eradicated when the result of 13C/14C-urea breath test goes from positive to negative
Gastrin-17 (pg/ml) | At baseline and 12, 26, 52 and 104 weeks
  To test the effects of Ho uGu Mi Xi on gastric function
Pepsinogen I (ng/ml) | At baseline and 12, 26, 52 and 104 weeks
  To test the effects of Ho uGu Mi Xi on gastric function
Pepsinogen II (ng/ml) | At baseline and 12, 26, 52 and 104 weeks
  To test the effects of Ho uGu Mi Xi on gastric function
Body weight (kg) | At baseline and 12, 26, and 52 weeks
  To test the regulating effect of Hou Gu Mi Xi on body weight
Body mass index (kg/m^2) | At baseline and 12, 26, and 52 weeks
  To test the regulating effect of Hou Gu Mi Xi on body weight.
Adverse events | At 6, 12, 26, 52 and 104 weeks
  Incidence of any adverse events. Safety outcome.
Severe adverse events | At 6, 12, 26, 52 and 104 weeks
  Incidence of any severe adverse events. Safety outcome.
Drug-related adverse events | At 6, 12, 26, and 52 weeks
  Incidence of any drug-related adverse events. Safety outcome.
Withdrawn due to adverse events | At 6, 12, 26, 52 and 104 weeks
  Incidence of any drug-related adverse events. Safety outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Zhu, Ph.D., Study Chair — Jiangxi University of Traditional Chinese Medicine
Locations (1):
- Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laine L, Jensen DM. Management of patients with ulcer bleeding. Am J Gastroenterol. 2012 Mar;107(3):345-60; quiz 361. doi: 10.1038/ajg.2011.480. Epub 2012 Feb 7. PMID 22310222
- [Background] Li Z, Zou D, Ma X, Chen J, Shi X, Gong Y, Man X, Gao L, Zhao Y, Wang R, Yan X, Dent J, Sung JJ, Wernersson B, Johansson S, Liu W, He J. Epidemiology of peptic ulcer disease: endoscopic results of the systematic investigation of gastrointestinal disease in China. Am J Gastroenterol. 2010 Dec;105(12):2570-7. doi: 10.1038/ajg.2010.324. Epub 2010 Aug 24. PMID 20736940
- [Background] Mohammadi M, Kashani SS, Garoosi YT, Tazehkand SJ. In vivo measurement of Helicobacter pylori infection. Methods Mol Biol. 2012;921:239-56. doi: 10.1007/978-1-62703-005-2_26. PMID 23015509
- [Background] Lanza FL, Chan FK, Quigley EM; Practice Parameters Committee of the American College of Gastroenterology. Guidelines for prevention of NSAID-related ulcer complications. Am J Gastroenterol. 2009 Mar;104(3):728-38. doi: 10.1038/ajg.2009.115. Epub 2009 Feb 24. PMID 19240698
- [Background] O'Connor A, Vaira D, Gisbert JP, O'Morain C. Treatment of Helicobacter pylori infection 2014. Helicobacter. 2014 Sep;19 Suppl 1:38-45. doi: 10.1111/hel.12163. PMID 25167944
- [Derived] Chen X, Yan D, Fang J, Liu W, Nie H, Lv N, Fang N, Gong J, Yu J, Jiang Y, Liu Z, Gan H, Fu Y, Yang D, Xiong Y, Liu D, Chen M, Wang Y, Wang Y, Sun X, Zhou X, Zhu W. Efficacy and safety of Hou Gu Mi Xi for peptic ulcer diseases: Study protocol for a randomized controlled trial. Medicine (Baltimore). 2019 Jul;98(29):e16561. doi: 10.1097/MD.0000000000016561. PMID 31335741